CLINICAL TRIAL: NCT03560765
Title: Training in the Use of Smartphones and Tablets to Improve Quality of Life in Visual Impairment - Mobile Electronic Devices for Visual Impairment
Brief Title: Mobile Electronic Devices for Visual Impairment
Acronym: MED4VI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer able to recruit due to COVID lockdowns
Sponsor: University of Manchester (Other)
Collaborators: City, University of London (Other); Schepens Eye Research Institute (Other)
Responsible Party: Principal Investigator, Chris Dickinson, Professor of Clinical Optometry, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5049/5050
Record Dates: First submitted 2018-05-22; First posted 2018-06-18 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Vision, Low
Keywords: Rehabilitation; Assistive technology
MeSH Terms: conditions — Vision, Low | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Using MED assigned buddy (Experimental): Participant has been randomly assigned a student volunteer buddy, and has chosen to purchase an MED following training
  Interventions: Device: MED; Other: Buddy
- Using MED training only (Active Comparator): Participant has been randomly assigned to not have a student volunteer buddy, and has chosen to purchase an MED following training
  Interventions: Device: MED
- No MED, assigned buddy (Active Comparator): Participant has been randomly assigned a student volunteer buddy, and has chosen not to purchase an MED following training
  Interventions: Other: Buddy
- No MED, no buddy (No Intervention): Participant has been randomly assigned to not have a student volunteer buddy, and has chosen not to purchase an MED following training

INTERVENTIONS:
Device: MED — Training in the use of mainstream electronic devices with accessibility options
  Other Names: smartphone; tablet; mobile electronic device
  Arms: Using MED assigned buddy; Using MED training only
Other: Buddy — A buddy who will meet with the participant regularly for social interaction, and assistance with use of any MED purchased
  Other Names: Student volunteer
  Arms: No MED, assigned buddy; Using MED assigned buddy

SUMMARY:
Mobile electronic devices (MED) including, smartphones and tablets, offer a new type of assistive technology for visually-impaired people (VIP). They offer the possibility to replace optical magnifiers for those with mild impairment, and braille or auditory for those with severe visual loss, using standard consumer devices, which are relatively cheap and convenient. However not all VIP and rehabilitation professionals are familiar with the devices and their potential.

In this study VIP who are interested in purchasing a MED will be recruited and trained. The effectiveness of this training will be determined by assessing the usage of devices by the participants from completion of training to 6 months, using questionnaires, and by remote monitoring of their MED. Validated questionnaires will be used to measure changes in quality of life, depression, adaptation to vision loss, and ability to carry out everyday tasks, before and after training, and 6 months later. Ongoing support has been found to be important when introducing users to new technology, in the form of volunteers to provide assistance and advice. The standard "training course only" model will therefore be compared to a scheme in which each participant is paired with a "buddy" (a university student) who can provide continuing support by visiting the VIP regularly at home.

DETAILED DESCRIPTION:
By converting text into speech and being cheaply and readily available, smartphones and tablets offer a completely new type of assistive technology for visually-impaired people (VIP). Research on these mobile electronic devices (MED) is relevant to rehabilitation and enablement of individuals with all types of visual impairment, with all degrees of severity. The majority of UK adults have a smartphone, but take-up is least amongst the over 75s who form the majority of the VI population. This is the population in whom MED have the greatest potential to reduce social isolation and increase independence, so it is important that the potential benefits are not restricted to those already comfortable with technology. Despite the great interest regarding what could be achieved with MED, evidence is currently lacking that they do provide significant improvements in quality of life, and that the specific training which is currently offered by many different organisations can help to facilitate effective use of MED.

The study aim is to evaluate the effectiveness of two different models of training in giving the user on-going access and improved quality of life. The two models to be compared will be a "training course only", versus a scheme in which each participant is paired with a "buddy" (a local university student) who can provide continuing assistance by visiting the participant at home.

VIP who are interested in purchasing a MED will be recruited and trained. The usage of devices will be assessed by questionnaire from completion of training to 6 months and through a tracking app. Validated questionnaires will be used to measure changes in quality of life, depression, adaptation to vision loss, and ability to carry out everyday tasks, before and after training, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* EITHER expresses an interest/referred specifically for MED training
* OR After evaluation it appears that MED would meet some/all requirements
* Willing to delay involvement in other forms of training or befriending for 6 months
* Has some form vision - does not rely exclusively on other senses
* Willing to travel for training/evaluation/meeting with buddy
* Agree not to seek additional formal/organised MED training elsewhere during the study
* Willing to fund any required MED personally
* Habitual language English
* 6 item Cognitive Impairment Test score 7 or lower
* Best corrected visual acuity logMAR 0.5 - 1.6 and/or log contrast sensitivity <1.2

Exclusion Criteria:

* Will be undergoing other one-to-one/group training (for anything) at the same time
* Will be undergoing other MED/general computer training at the same time
* Will be actively enrolled in a new befriending/social group
* Already knows basics of MED and wants training on advanced skills
* Obvious cognitive impairment or uncorrected hearing loss such that communication is through a third party
* If updated Rx would improve VA by 2 lines or more, participant should be recommended to seek eye exam and then be re-evaluated 1 month later
* Visual condition likely to be treated/improved within study period such that MED no longer required

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Vision QoL Core Measure VCM-1 | 2 months
  A 9-item instrument to measure vision related quality of life. Each item scored from 0-4 with a maximum score of 36. Low score represents poor QoL.
Vision QoL Core Measure VCM-1 | 6 months
  A 9-item instrument to measure vision related quality of life. Each item scored from 0-4 with a maximum score of 36. Low score represents poor QoL.

SECONDARY OUTCOMES:
Centre for Epidemiological Studies Depression Scale (CES-D) | 2 months
  A 20-item instrument to measure self-reported depression. Each item scored from 0-3 with a maximum score of 60. Low score represents an absence of depression.
Centre for Epidemiological Studies Depression Scale (CES-D) | 6 months
  A 20-item instrument to measure self-reported depression. Each item scored from 0-3 with a maximum score of 60. Low score represents an absence of depression.
Acceptance and Self Worth Adjustment Scale ASWAS | 2 months
  A 19-item instrument which measures adaptation to acquired visual loss. Questions relate to self-esteem, attitudes, acceptance, self-efficacy, and locus of control. Each item scored from 0-4, and maximum score of 76 represents good acceptance and self-worth.
Acceptance and Self Worth Adjustment Scale ASWAS | 6 months
  A 19-item instrument which measures adaptation to acquired visual loss. Questions relate to self-esteem, attitudes, acceptance, self-efficacy, and locus of control. Each item scored from 0-4, and maximum score of 76 represents good acceptance and self-worth.
Modified Manchester Low Vision Questionnaire with Canadian Occupational Performance Measure | 2 months
  A questionnaire in 3 sections, each of which are independent.. Section 1 describes how the participant carries out a list of everyday activities (with which assistive device, and with how much assistance). Section 2 grades the amount of time that different aids are used (graded fro 0-4 with 4 representing the most usage). In Section 3 the participant identifies 5 activities which they would like to improve, and grades on a scale of 0-10) the importance of the task, their performance, and their satisfaction with their performance of it. An "importance x satisfaction" and "importance x performance" score for each activity are calculated.
Modified Manchester Low Vision Questionnaire with Canadian Occupational Performance Measure | 6 months
  A questionnaire in 3 sections, each of which are independent. Section 1 describes how the participant carries out a list of everyday activities (with which assistive device, and with how much assistance). Section 2 grades the amount of time that different aids are used (graded fro 0-4 with 4 representing the most usage). In Section 3 the participant identifies 5 activities which they would like to improve, and grades on a scale of 0-10) the importance of the task, their performance, and their satisfaction with their performance of it. An "importance x satisfaction" and "importance x performance" score for each activity are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Dickinson, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - City University of London, London
  - University of Manchester, Manchester